CLINICAL TRIAL: NCT06357832
Title: A Prospective, Randomized, Controlled, Multicenter Trial to Evaluate the Safety and Efficacy of Deep Transcranial Magnetic Stimulation (Deep TMS) With a New Stimulation Protocol in Subjects With Major Depression Disorder (MDD)
Brief Title: New Investigational Stimulation Protocol for Treatment of Major Depression Disorder (MDD)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTP-ACCiTBS-00
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Investigational stimulation group (Experimental): The experimental group will receive the new investigational deep TMS protocol
  Interventions: Device: Brainsway Deep TMS System
- Standard-of-care stimulation group (Active Comparator): The control group will receive the currently FDA-cleared standard-of-care deep TMS protocol.
  Interventions: Device: Brainsway Deep TMS System

INTERVENTIONS:
Device: Brainsway Deep TMS System — The BrainsWay Deep TMS device is intended for the treatment of depressive episodes in patients suffering from Major Depressive Disorder (MDD). The device technology is based on the application of deep brain TMS by means of repetitive pulse trains at a determined frequency.
  Other Names: Brainsway Deep TMS Device

SUMMARY:
The BrainsWay Deep Transcranial Magnetic Stimulation (Depp TMS) device is intended for the treatment of depressive episodes in patients suffering from Major Depressive Disorder (MDD). The device technology is based on the application of deep brain TMS by means of repetitive pulse trains at a determined frequency. The purpose of the current study is to evaluate the safety and effectiveness of a new investigational stimulation protocol delivered with the BrainsWay Deep TMS device, for the treatment of MDD, demonstrating that it is non-inferior to the current standard-of-care stimulation protocol, in a randomized, controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients.
* Men and women 22-68 years of age.
* Primary Diagnostic and Statistical Manual (DSM-V) diagnosis of Major Depression, single or recurrent episode confirmed by the Quick Structured Clinical Interview for the DSM-5 Disorders (QuickSCID-5), with the additional requirements of a current episode ≥4 weeks and CGI-S ≥4.
* Current depressive episode is less than 5 years in duration (the definition of an episode is demarcated by a period of ≥2 months in which the patient did not meet full criteria for the DSM-V definition of major depressive episode);
* Total HDRS-21 ≥20 and Item 1 score ≥2 at the screening visit;
* The patient did not respond to at least one antidepressant treatment, i.e., a minimum of 1 and a maximum of 4 antidepressant drug trials, of adequate dose and duration (defined as a minimum level of 3 on the Antidepressant Treatment History Form - Short Form (ATHF-SF)) in the current episode; or Patients who have not completed antidepressant trials of adequate dose and duration (defined as a level of 1-2 on the ATHF-SF) due to intolerance to therapy, if they have demonstrated intolerance to 2 or more antidepressant medications in the current episode.
* Capable and willing to provide informed consent
* Able to adhere to the treatment schedule.
* Patient is stable on medication for 2 month and is not expected to change medication during the study period.
* Satisfactory safety screening questionnaire for transcranial magnetic stimulation.

Exclusion Criteria:

* Investigators, site personnel directly affiliated with this study, and their immediate families (immediate family is defined as a spouse, parent, child or sibling, whether by birth or legal adoption);
* Individuals diagnosed by the Investigator with the following conditions (current unless otherwise stated):
* Depression secondary to a general medical condition, or substance-induced;
* Substance abuse disorder within the past 3 months (except nicotine and caffeine). Note that use of cannabis for medical reasons in a stable regimen is permitted as long as the investigator excludes abuse of the substance.
* Any psychotic disorder (lifetime), including schizoaffective disorder or major depression with psychotic features or Bipolar disorder.
* Post-traumatic stress disorder (current or within the past year)
* Current (within 12 months of baseline) generalized anxiety disorder, panic disorder or social anxiety disorder as assessed by the investigator to be primary, causing a higher degree of distress or impairment than MDD.
* Presence (within 12 months of baseline) of a personality disorder (such as antisocial, schizotypal, histrionic, borderline, narcissistic) as assessed by the investigator to be primary, causing a higher degree of distress or impairment than MDD.
* Individuals with a significant neurological disorder or insult including (but not limited to):
* Any condition likely to be associated with increased intracranial pressure
* Space occupying brain lesion
* Any history of seizure EXCEPT those therapeutically induced by Electroconvulsive T Therapy (ECT) or febrile seizures
* History of cerebrovascular accident
* Transient ischemic attack within two years
* Cerebral aneurysm
* Dementia
* Mini Mental State Exam score of less than or equal to 24
* Parkinson's disease
* Huntington's chorea
* Multiple sclerosis
* Individuals with a first-degree relative family history of seizure.
* ECT treatment within 3 months prior to the screening visit
* History of treatment with Vagus Nerve Stimulation (VNS)
* History of treatment with Deep Brain Stimulation (DBS)
* Use of any investigational drug within 4 weeks of the baseline visit
* Present suicidal risk as assessed by the investigator or significant suicide risk based on HDRS-21 item 3 score of 3 or 4, or significant suicide risk as assessed using the Scale for Suicide Ideation (SSI), or a history of attempted suicide in the last year.
* Any self-inflicted harm in the past 3 months not in the context of suicidal ideation.
* Conductive, ferromagnetic or other magnetic-sensitive metals implanted in the head (excluding the mouth) or within 10 cm of the treatment coil (e.g., cochlear implants, implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, shrapnel, surgical clips, fragments from welding or metal work).
* Individuals who have cardiac pacemakers or active implantable electrodes/neurostimulators within 30 cm of the treatment coil.
* If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the rTMS trial
* Clinically significant medical condition in the opinion of the Investigator.
* Known or suspected pregnancy
* Women who are breast-feeding
* Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.

Ages: 22 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HDRS)-21 score in the investigational group | 6 weeks
  Change in Hamilton Depression Rating Scale (HDRS)-21 scores from baseline to the 6 week follow up

SECONDARY OUTCOMES:
Response rate in the investigational group | 6 weeks
  The percentage of patients in the treatment group who had a reduction of ≥50% in HDRS-21 score from baseline to the 6 week follow up
Remission rate in the investigational group | 6 weeks
  The percentage of patients in the investigational group with an HDRS-21 score < 10 at 6 weeks
Change in Clinical Global Impression-Severity (CGI-S) scores in the investigational group | 6 week
  Change in Clinical Global Impression-Severity (CGI-S) scores from baseline to the 6 week follow up
Change in Clinical Global Impression Improvement (CGI-I) scores in the investigational group | 6 week
  Change in Clinical Global Impression Improvement (CGI-I) scores from baseline to the 6 week follow up

CONTACTS AND LOCATIONS:
Locations (9):
- United States (7):
  - Novus Neurology, Tuscaloosa, Alabama
  - Inland Psychiatric Medical Group, Inc., Redlands, California
  - DTMS Center LLC, Palm Beach, Florida
  - Fermata Health, Brooklyn, New York
  - Complete Mind Care of PA, Abington, Pennsylvania
  - ClearPath Psychiatry, Seattle, Washington
  - PsyCare, South Charleston, West Virginia
- Asha Neuromodulation Clinic, Hyderabad, Telangana, India
- Be'er Ya'aqov-Ness Ziona Mental Health Center, Be’er Ya‘aqov, Israel